CLINICAL TRIAL: NCT03481985
Title: The Effect of Fontan Fenestration Closure on Hepatic Stiffness
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Rahul Rathod, Cardiologist, Boston Children's Hospital
Other Study IDs: IRB-P00027110
Record Dates: First submitted 2018-03-07; First posted 2018-03-29 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Single-ventricle; Hepatic Congestion
Keywords: Fontan-associated liver disease
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Other: Fenestration status — The exposure variable will be status of the Fontan fenestration

SUMMARY:
The overarching goal of this project is to discern how closure of Fontan fenestrations in patients with single ventricle heart disease will affect hepatic congestion, a major determinant of chronic liver disease. We will employ transient elastography (Fibroscan) to obtain liver stiffness measurements (LSM) before and after fenestration closure to study the impact of this intervention on hepatic congestion.

DETAILED DESCRIPTION:
Methods Eligible patients will be contacted in advance of hospitalization for catheterized fenestration closure to introduce goals of study and review risks and benefits of participation. At the time of catheterization, the study objectives and consent forms will be explained, allowing sufficient time for questions. To ensure full comprehension of the study, the parent or guardian will be asked to describe his or her participation in the trial.

Using the Fibroscan (Echosens, Paris, France), a transient elastography device, a liver stiffness measurement (LSM) will be obtained prior to the catheterization. On the post-catheterization day, a repeat measurement will be obtained. Transient elastography will be performed by trained study investigators who were certified by the manufacturer.

To obtain an LSM, the appropriate-sized Fibroscan probe must be selected and then aimed in the right upper quadrant space through an intercostal space. For patients with heterotaxy or situs inversus, adjustments in probe positioning may be needed to obtain reliable measurement. Probe selection (small, medium, or large) will be directed by manufacturer guidelines, based on thoracic perimeter.

The operator is guided by an image to locate an appropriate section of liver. The Fibroscan device transmits an elastic shear wave through the hepatic parenchyma and then measures the propagation of the wave through a known distance of liver tissue to calculate a transmission velocity. Using the shear velocity and the mass density of the liver parenchyma, the principles of Young's modulus are invoked to estimate the Elasticity of the tissue. The elasticity is summarized as a liver stiffness measurement (LSM), which is a continuous variable that is reported in kilopascals (kPa). Each LSM outcome value is based on a minimum of ten valid assessments measured in succession. The validity of each individual measurement is determined by the device and the interquartile range of the measurements should fall within 30% of the median LSM. The Fibroscan data collection method is non-invasive and efficient. LSM will be obtained after fasting for a minimum of three hours and without administration of sedating agents/anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Functional Single ventricle patients after a fenestrated lateral tunnel or extra-cardiac Fontan
* Patients scheduled for possible fenestration closure in the catheterization laboratory
* Informed consent has been obtained

Exclusion Criteria:

* Patients with spontaneous closure of Fenestration
* Ascites
* Ventilatory requirement
* Implantable cardiac device
* Ongoing inotropic support
* Pregnancy
* Inability to tolerate four hour pre-procedure fasting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any functional single-ventricle patients undergoing catheterization for Fontan fenestration closure will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Immediate change in liver stiffness | Patients will have measurements on day of catheterization and day after catheterization. They will be followed through study completion, an average of 6 months.
  Immediate change in Liver stiffness measurement (measured by Transient Elastography)he first measurement will be obtained on the day of the catheterization (for fenestration closure). The second measurement will be post-fenestration closure and will be obtained on the day after the catheterization.

SECONDARY OUTCOMES:
Short term change in liver stiffness | The first measurement will be obtained on the day of the catheterization (for fenestration closure). The long-term outcome measurement will be obtained three months afterwards. They will be followed through study completion, an average of 6 months.
  Short term change in Liver stiffness measurement (measured by Transient Elastography). The first measurement will be obtained on the day of the catheterization (for fenestration closure). The long-term outcome measurement will be obtained three months after the catheterization procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Rathod, MD, Principal Investigator — Cardiologist/Principal Investigator
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No